CLINICAL TRIAL: NCT05284656
Title: The Potential Nephro-protective Effect of Folic Acid and/or Pentoxifylline on Patients With Chronic Kidney Disease
Brief Title: Effect of Folic Acid and/or Pentoxifylline on Patients With Chronic Kidney Disease
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Amira Reda Muhammad Galal, Principal investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interventional
Record Dates: First submitted 2022-02-16; First posted 2022-03-17 (Actual); Results first posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Folic Acid; Pentoxifylline

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- folic acid Group (Experimental): 20 patients will receive folic acid 500 µg per day with their standard therapy for 6 months.
  Interventions: Drug: folic acid
- Pentoxifylline Group (Experimental): 20 patients will receive Pentoxifylline ( TRENTAL® Tablets, 400 mg) twice daily with their standard therapy for 6 months.
  Interventions: Drug: Pentoxifylline 400 MG
- folic acid and pentoxifylline Group (Experimental): 20 patients will receive combination therapy of folic acid5 mg per day and pentoxifylline ( TRENTAL® Tablets, 400 mg) twice daily with their standard therapy for 6 months
  Interventions: Drug: combination of Pentoxifylline 400 MG and Folic Acid
- control group (No Intervention): 20 patients will receive their standard therapy only.

INTERVENTIONS:
Drug: combination of Pentoxifylline 400 MG and Folic Acid — drugs used to delay progression of chronic kidney disease
  Other Names: combination of Trental SR 400mg and Folic acid
  Arms: folic acid and pentoxifylline Group
Drug: folic acid — drugs used to delay progression of chronic kidney disease
  Arms: folic acid Group
Drug: Pentoxifylline 400 MG — drugs used to delay progression of chronic kidney disease
  Other Names: Trental SR 400mg
  Arms: Pentoxifylline Group

SUMMARY:
The aim of this study is to evaluate the effect of administration of folic acid and /or pentoxifylline on patients with chronic kidney disease (CKD).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a worldwide public health problem, with adverse outcomes of kidney failure, cardiovascular disease (CVD), and premature death. Chronic kidney disease (CKD) affects between 8% and 16% of the population worldwide.Defined by a glomerular filtration rate (GFR) of less than 60 mL/min/1.73 m2, albuminuria of at least 30 mg per 24 hours, or markers of kidney damage (eg, hematuria or structural abnormalities such as polycystic or dysplastic kidneys) persisting for more than 3 months.That nutrient loss because of diet restriction and chronic inflammation contributed by CKD itself may stimulate progression in advanced chronic kidney disease. Folic acid was then selected as a nutrient intervention. In the mean time, pentoxifylline was well studied in this field for its anti-inflammatory effects.Pentoxifylline (PTF) appears to improve circulation through its ability to alter erythrocyte deformability and enhances capillary microcirculation. This hemorheological property and the potential capacity in decreasing intraglomerular pressure has led to recent interest in PTF as a therapeutic agent in patients with kidney disease. In addition to these properties, PTF has an effect on inflammation, oxidative stress and endothelial function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have chronic kidney disease(CKD) stages 3-5
2. Aged between18 - 60 years old.
3. Both sexes.
4. Stable clinical condition defined as no hospitalizations or cardiovascular events within the 3 months before screening
5. Stable renal function (baseline serum creatinine had to have not increased by 50% in the 3 months before screening)
6. No changes in concomitant medication during the study.
7. Patients who accept to participate in the study.

Exclusion Criteria:

1. Pregnant women
2. Current use of PTF
3. Contraindication to use of PTF drug: history of PTF or theophylline allergy, history of severe retinal hemorrhage or recent cerebral hemorrhage
4. Those with active infections or inflammatory diseases or HIV infection
5. Those with chronic liver disease .
6. Patients who had received immunosuppressive therapy
7. Non-compliant patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-01-08 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-12-19 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab AlKasaby, Principal Investigator — Professor and Head of Clinical Pharmacy Department, Faculty of Pharmacy (Girls), Al-Azhar University
Locations (1):
- Al Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Galal ARM, Teama NM, Abu-Elfotuha K, Alatawi AD, Alshareef H, Hamdan AME, Aljabri A, Alshibani M, Zalat ZAM. The potential adding therapeutic effect of pentoxifylline and/or folic acid for chronic kidney disease patients: randomized controlled trial. BMC Nephrol. 2025 Aug 18;26(1):468. doi: 10.1186/s12882-025-04399-3. PMID 40826392

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: some patient are excluded from the study as they donnot meet the inclusion criteria
Period: Overall Study
Arm/Group | Folic Acid Group | Pentoxifylline Group | Folic Acid and Pentoxifylline Group | Control Group
Started | 20 | 20 | 20 | 20
Completed | 20 | 20 | 20 | 20
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Folic Acid Group | Folic Acid and Pentoxifylline Group | Pentoxifylline Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.25 (6.64) | 51.80 (6.7) | 52.20 (7.2) | 51.6 (6.6) | 51.96 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 10 | 12 | 53
  Male | 5 | 4 | 10 | 8 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
glomular filtration rate [Mean (Standard Deviation); unit: ml/min] — glomular filtration rate is measured from serum creatinine to measure kidney function
  ml/min | 22.15 (11.12) | 17.25 (7.217) | 17.85 (8.6) | 21.87 (9.7) | 19.78 (9.15)

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Creatinine Level
Description: Change was calculated as the value at 6 months minus the value at baseline.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Folic Acid Group | Pentoxifylline Group | Folic Acid and Pentoxifylline Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20 | 20
mg/dl | 3.118 (1.203) | 3.335 (1.149) | 3.535 (0.9109) | 2.872 (0.8901)

2. Secondary Outcome: Serum Ferritin in ng/ml
Description: increase in serum ferritin from baseline
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Folic Acid Group | Pentoxifylline Group | Folic Acid and Pentoxifylline Group | Control Group
Number analyzed (Participants) | 20 | 20 | 20 | 20
ng/ml | 200.6 (66.18) | 334.1 (230.2) | 245.1 (115.7) | 235.3 (185.1)

3. Other Pre Specified Outcome: Protein/ Creatinine Ratio(P/C) (mg Protein/mg Creatinine)
Description: change in Protein/ creatinine ratio for determination of proteinuria
Time Frame: 6 months
Reporting Status: Not Posted, anticipated posting 2025-12

ADVERSE EVENTS:
Time Frame: patient are followed up for 6 months for any adverse events
Description: the drug is safe and approved by FDA and the assessment of adverse event was collected based on weekly questionnaire
Arm/Group | Folic Acid Group | Pentoxifylline Group | Folic Acid and Pentoxifylline Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/56/NCT05284656/Prot_000.pdf